CLINICAL TRIAL: NCT05241899
Title: A Multicenter, Open Label，Single Arm，Phase II Study to Evaluate the Effect and Safety Fruquintinib Combined With RC48 in the Treatment of Previously Treated HER2-positive Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (G/GEJ) Cancer
Brief Title: A Phase II Clinical Study of Fruquintinib Combined With RC48 in the Treatment of Previously Treated HER2-positive Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (G/GEJ) Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013
Record Dates: First submitted 2022-02-06; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer
Keywords: Fruquintinib，RC48，G/GEJ cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; RC48 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib + RC48 (Experimental): Fruquintinib + RC48
  Interventions: Drug: Fruquintinib + RC48

INTERVENTIONS:
Drug: Fruquintinib + RC48 — Fruquintinib (4mg orally, once daily for 3 wks on/1 wk off) combined with of RC48( 2.5mg/kg by intravenous infusion during 30-90 min every 2 weeks)

SUMMARY:
Although Pembrolizumab plus trastuzumab and chemotherapy is the standard of care for first-line treatment of HER2-positive advanced or metastatic gastric or gastroesophageal junction (G/GEJ) cancer,there is no established therapy in the second-line setting.

RC48 showed promising activity with manageable safety in patients with HER2-overexpressing, advanced G/GEJ cancer who have previously received at least two lines of chemotherapy.Fruquintinib in combination with Paclitaxel demonstrated encouraging preliminary clinical antitumor activity in patients with advanced GC in ph1b/2 study.

This study is aimed to evaluate the efficacy and safety of Fruquintinib in combination with RC48 in the treatment of previously treated HER2-positive locally advanced or metastatic gastric or gastroesophageal junction (G/GEJ) cancer.

DETAILED DESCRIPTION:
This study is a phase II, single arm study with main purpose to evaluate the safety, tolerability and efficacy of Fruquintinib in combination with RC48 in the treatment of previously treated HER2-positive locally advanced or metastatic gastric or gastroesophageal junction (G/GEJ) cancer.

All eligible patients received Fruquintinib (4mg orally, once daily for 3 wks on/1 wk off) combined with of RC48( 2.5mg/kg by intravenous infusion during 30-90 min every 2 weeks) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75years (inclusive);
2. Body weight ≥40 kg;
3. Physical status score (ECOG score) 0-1;
4. Expected survival >12 weeks.;
5. At least one measurable lesion (according to RECIST1.1);
6. Histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic HER2 positive G/GEJ cancer;
7. HER2-positive defined as either immunohistochemistry (IHC) 3+ or IHC 2+ in combination with in-situ hybridization positive (ISH+) or fluorescent in-situ hybridization (FISH), as assessed by central review on primary or metastatic tumor;
8. Fail in previous first-line standard chemotherapy;
9. prior therapy does not need to have included a HER2-directed therapy;
10. Adjuvant or neoadjuvant therapy for AGC is allowed.
11. Absence of major post-operative complications or other clinical conditions that, in the opinion of the investigator, would contraindicate adjuvant chemotherapy 8. Adequate hematological function defined by absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet count ≥100 × 109/L, and hemoglobin ≥9 g/dL (blood transfusion before recruitment is allowed)
12. Adequate hepatic function defined by a total bilirubin level ≤1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤2.5 × ULN 10. Adequate renal function defined by an estimated creatinine clearance ≥30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) 11. Negative serum or urine pregnancy test at screening for women of childbearing potential 12. Fertile men and women must agree to take highly effective contraceptive precautions during, and for 6 months after the last dose of chemotherapy or for 1 month after the last dose of Tislelizumab

Exclusion Criteria:

1. An interval shorter than 21 days from the last dose of chemotherapy or HER2-directed therapy until the time of randomization
2. Prior treatment with RC48, Fruquintinib, or apatinib either as single agents or as part of a treatment regimen.
3. Treatment with any investigational anticancer drug within 21 days of the first study treatment administration
4. More than one prior line of therapy for advanced G/GEJ cancer;
5. History of other malignancy within the previous 5 years except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other malignancies with an expected curative outcome
6. Brain metastases that are untreated or symptomatic or require any radiation, surgery, or steroid therapy to control symptoms from brain metastases within 1 month of randomization
7. Peripheral neuropathy Grade >/=2
8. Uncontrolled cardiopulmonary dysfunction (e.g., high blood pressure, serious cardiac arrhythmia)
9. Other current, severe, uncontrolled systemic disease (e.g., clinically significant metabolic disease, wound healing disorders, ulcers)
10. Clinically significant bleeding within 30 days before enrollment
11. For female participants, current pregnancy or lactation
12. Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
13. Infection with Human immunodeficiency virus (HIV) or hepatitis B virus, hepatitis C virus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-05-07 (Estimated); Primary Completion 2023-05-07 (Estimated); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | from randomization until death due to any cause, assessed up to 3 year
  every two months follow up after EOT observation period at 30 days after the last medication
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China